CLINICAL TRIAL: NCT03827590
Title: Phase III Clinical Trials to Assess the Efficacy and Safety of HLIM for Symptomatic Relief of Cough and Sputum in Patients With Acute Upper Respiratory Tract Infection or Acute Bronchitis
Brief Title: Clinical Trials to Assess the Efficacy and Safety of HLIM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SamA Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HLIM(SA16002)
Record Dates: First submitted 2019-01-10; First posted 2019-02-01 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Acute Upper Respiratory Tract Infection; Acute Bronchitis
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- HLIM (Experimental): HLIM+SA160021 Placebo+SA160022 Placebo
  Interventions: Drug: Test
- SA160021 (Active Comparator): HLIM Placebo+SA160021+SA160022 Placebo
  Interventions: Drug: Active Comparator Control 1
- SA160022 (Active Comparator): HLIM Placebo+SA160021 Placebo+SA160022
  Interventions: Drug: Active Comparator Control 2
- Placebo (Placebo Comparator): HLIM Placebo+SA160021 Placebo+SA160022 Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Test — three times a day for five days
  Other Names: HLIM+SA160021 Placebo+SA160022 Placebo
  Arms: HLIM
Drug: Active Comparator Control 1 — three times a day for five days
  Other Names: HLIM Placebo+SA160021+SA160022 Placebo
  Arms: SA160021
Drug: Active Comparator Control 2 — three times a day for five days
  Other Names: HLIM Placebo+SA160021 Placebo+SA160022
  Arms: SA160022
Drug: Placebo — three times a day for five days
  Other Names: HLIM Placebo+SA160021 Placebo+SA160022 Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of HLIM

DETAILED DESCRIPTION:
A randomized, double-blind, active-controlled, multicenter phase 3 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 and 75
* Weight more than 11.5 kg

Exclusion Criteria:

* Has a history of hypersensitivity to IP ingredients
* Hypertension or Diabetes
* Smoking more than 20 pack-years

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 487 (Estimated)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in BSS(Bronchitis Severity Score)-cough domain of active comparator control 2 versus placebo | 5 days
  0(absent) ~ 4(very severe), Total Score: 0~20
Changes in BSS(Bronchitis Severity Score) total score of each active comparator control group compared to the test group | 5 days
  0(absent) ~ 4(very severe), Total Score: 0~20

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, Guro-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided